CLINICAL TRIAL: NCT07307599
Title: Optimizing Fluid Resuscitation in Adults With Major Burns: A Randomized Trial of Burn Navigator™ Versus Parkland Formula
Acronym: FLARE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alnas Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Abdel hafiez, Head of Burn ICU, Alnas Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHDIRB-NA-240823-01UC-NPO-N020
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Resuscitation, Burn
Keywords: resuscitation; burn, 2nd degree; burn, 3rd degree; Burn; Severe burn; critically ill; Golden hours
MeSH Terms: conditions — Burns; Critical Illness | interventions — Resuscitation; HES 130-0.4

STUDY DESIGN:
Intervention Model Description: This study uses a two-group comparative design to evaluate fluid resuscitation strategies in adult burn patients. Participants will be allocated into two parallel groups. The control group will receive fluid resuscitation guided by the standard Parkland formula during the first 48 hours post-burn. The intervention group will receive fluid resuscitation directed by the Burn Navigator™ system, which provides hourly recommendations based on patient-specific variables including urinary output, weight, burn size, and time post-injury. Both groups will be monitored for adequacy of resuscitation, complications of under- or over-resuscitation, and overall clinical outcomes.
Who Masked: Participant
Masking Description: This study will use a single-blind parallel design in which participants are unaware of the resuscitation method assigned to them. Clinical staff delivering care will know the allocation in order to administer either the Parkland formula or the Burn Navigator™-guided regimen; however, participants will not be informed of which fluid management strategy they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkland Arm (Active Comparator): Participants in this arm will receive fluid resuscitation according to the conventional Parkland formula, which recommends 4 mL/kg/TBSA of crystalloid fluids during the first 24 hours post-burn. Half of the calculated volume will be administered in the first 8 hours after injury, with the remainder given over the next 16 hours. Adjustments may be made based on clinical response, including urine output and hemodynamic status. This approach represents the standard of care for initial burn resuscitation and will be used as the comparator for evaluating the effectiveness of Burn Navigator™-guided resuscitation.
  Interventions: Other: Resuscitation (Voluven)
- Burn Navigator Arm (Experimental): Participants in this arm will receive fluid resuscitation guided by the Burn Navigator™ decision-support system. This software uses real-time mathematical modeling based on weight, burn size, time post-injury, prior fluid infusion, and the last three urine output measurements to generate hourly recommended fluid rates. The goal is to optimize resuscitation, avoid over- or under-resuscitation, and maintain adequate end-organ perfusion during the first 48-72 hours post-burn. Clinical teams will follow the system's recommendations unless medically contraindicated.
  Interventions: Device: Burn Navigator

INTERVENTIONS:
Device: Burn Navigator — Participants in this arm will receive fluid resuscitation guided by the Burn Navigator™ decision-support system. This software uses real-time mathematical modeling based on weight, burn size, time post-injury, prior fluid infusion, and the last three urine output measurements to generate hourly recommended fluid rates. The goal is to optimize resuscitation, avoid over- or under-resuscitation, and maintain adequate end-organ perfusion during the first 48-72 hours post-burn. Clinical teams will follow the system's recommendations unless medically contraindicated.
  Arms: Burn Navigator Arm
Other: Resuscitation (Voluven) — Resuscitation ringer / Resuscitation (Voluven) + Plasma
  Arms: Parkland Arm

SUMMARY:
Burn injuries affecting ≥20% TBSA trigger major fluid shifts requiring aggressive fluid resuscitation to prevent burn shock. Traditional formulas such as the Parkland and Modified Brooke estimate initial 24-hour fluid needs, but both under- and over-resuscitation can cause serious complications. To improve accuracy, the Burn Navigator™ (BN) system uses patient-specific, real-time data and mathematical modeling to guide hourly fluid adjustments. Previous studies showed reduced fluid volumes compared to manual resuscitation, but comprehensive evaluation across settings is lacking.

This study aims to compare Burn Navigator™-guided resuscitation versus the conventional Parkland formula in adult burn patients during the first 24-72 hours post-injury, focusing on achieving optimal fluid balance and preventing complications.

DETAILED DESCRIPTION:
Burn injuries vary widely in cause and severity but share the fundamental pathologic feature of liquefactive necrosis of the skin, the body's largest organ and a key component of the immune defense system. When burns involve 20% or more of the total body surface area (TBSA), a profound systemic inflammatory response develops. This response causes extensive fluid shifts and third spacing, leading to loss of intravascular volume, reduced organ perfusion, and a high risk of burn shock. To counter these physiological changes, intravenous fluid resuscitation during the first 24-48 hours post-burn is an essential component of management.

Traditional burn resuscitation guidelines-most notably the Parkland formula (4 mL/kg/TBSA) and the Modified Brooke formula (2 mL/kg/TBSA)-provide initial estimates for required fluid volumes. However, these formulas are static and may not reflect rapid, patient-specific changes. Excessive fluid administration can result in life-threatening complications such as abdominal, extremity, or ocular compartment syndrome, while inadequate resuscitation can precipitate acute kidney injury, burn shock, or multi-organ failure.

Modern approaches emphasize dynamic hourly titration of fluids based on physiologic response, particularly urinary output (UO), to avoid under- and over-resuscitation. To support clinicians in making real-time adjustments, the Burn Resuscitation Decision Support System (BRDSS) was developed by the United States Army Institute of Surgical Research and UTMB. Now commercialized as the Burn Navigator™, this system uses a mathematical model incorporating UO trends, fluid infusion rates, burn size, body weight, and time post-injury to generate hourly fluid recommendations. Studies have shown it can reduce overall fluid exposure compared to manual adjustments.

Despite widespread adoption in military and civilian burn centers, there has been no comprehensive evaluation of its performance across varied clinical environments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Total Burn Surface Area (TBSA) ≥20%
* weight > 40 kg
* Informed consent provided

Exclusion Criteria:

* Primary electrical burn
* Pregnancy
* End-stage renal disease or decompensated heart failure
* Burns associated with trauma (polytrauma)
* Refusal or withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total fluid volume administered within the first 24 hours normalized to body weight and %TBSA | 24 hours
  Total fluid volume administered within the first 24 hours normalized to body weight and %TBSA

SECONDARY OUTCOMES:
Time to target urine output (in hours) | 48hours
  Time to target urine output (in hours)
Fluid creep occurrence (>6 ml/kg/%TBSA in first 24 hours ) | 24 Hours
  Pulmonary edema Abdominal or extremity compartment syndrome Shock

OTHER OUTCOMES:
30 day mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- ALNAS Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided